CLINICAL TRIAL: NCT04118387
Title: Central Sleep Apnea: Physiologic Mechanisms to Inform Treatment
Brief Title: Central Sleep Apnea : Physiologic Mechanisms to Inform Treatment
Acronym: CSA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NURR-001-19S; I01CX001944 (NIH)
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Sleep Disordered Breathing; Able Bodied
Keywords: Central sleep apnea; Polysomnography (PSG); Respiratory arousal threshold; Apnea Hypopnea index; Central Apnea Hypopnea Index; Breathing instability; Apneic Threshold (AT); Peripheral chemoreflex sensitivity; CO2 reserve; Plant gain; Controller gain
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Central | interventions — Acetazolamide; Zolpidem; Buspirone

STUDY DESIGN:
Intervention Model Description: Specific Aim (1) is to determine the effect of combination therapy aiming to dampen chemoreceptor sensitivity AND decreasing plant gain. We hypothesize that combined therapy with PAP, acetazolamide and oxygen will be superior to each intervention alone in reducing CAHI and the CO2 reserve during sleep in patients with central sleep apnea. Specific Aim (2) is to determine the effect of decreasing respiratory-related arousals on the propensity to develop central apnea. We hypothesize that administration of PAP and zolpidem, will decrease respiratory-related arousals, CAHI and the CO2 reserve during sleep in patients with CSA compared to placebo. Specific Aim (3) is to determine the effect of augmenting serotonin A1 receptor activity on breathing during sleep. We hypothesize that administration of PAP and buspirone, a serotonin A1 receptor agonist; will reduce the propensity to central apnea during sleep in Veterans with central sleep apnea.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- acetazolamide (Active Comparator): To determine the effect of dampening chemoreceptor sensitivity AND decreasing plant gain. The investigators hypothesize that combined therapy with PAP, acetazolamide and oxygen will be superior to PAP plus each intervention alone or placebo in reducing CAHI and the CO2 reserve during sleep in Veterans with CSA.
  Interventions: Drug: Acetazolamide + supplemental oxygen + PAP therapy
- zolpidem (Active Comparator): To determine the effect of decreasing respiratory-related arousals on the propensity to develop central apnea. The investigators hypothesize that administration of PAP and zolpidem, will decrease respiratory-related arousals, CAHI and the CO2 reserve during sleep in Veterans with CSA compared to PAP plus placebo.
  Interventions: Drug: Zolpidem + PAP therapy
- buspirone (Active Comparator): To determine the effect of augmenting serotonin A1 receptor activity on breathing during sleep. The investigators hypothesize that administration of PAP and buspirone, a serotonin A1 receptor agonist; will reduce the propensity to central apnea during sleep in Veterans with CSA compared to PAP plus placebo.
  Interventions: Drug: Buspirone + PAP therapy

INTERVENTIONS:
Drug: Acetazolamide + supplemental oxygen + PAP therapy — Every participant will undergo measurement of the apneic threshold. The apneic threshold (AT) can be determined by inducing central apnea using non-invasive ventilation (NIV) or eliminating central apnea using supplemental CO2. The requisite change to induce central apnea is referred to as the CO2 reserve, which can be positive or negative. The central apnea index and the apneic threshold will be measured while participants receiving medication or oxygen (or both). In addition, participants will get PAP therapy during all the conditions.
  Arms: acetazolamide
Drug: Zolpidem + PAP therapy — The central apnea index and the apneic threshold will be compared under two conditions: zolpidem or placebo. In addition, participants will get PAP therapy during both the conditions.
  Arms: zolpidem
Drug: Buspirone + PAP therapy — The central apnea index and the apneic threshold will be compared under two conditions: buspirone or placebo. In addition, participants will get PAP therapy during both the conditions.
  Arms: buspirone

SUMMARY:
Central sleep apnea (CSA) is common in patients with heart failure and those using opioid analgesics. Unfortunately, effective treatment of central apnea remains elusive, pressure therapy given the modest efficiency of positive airway pressure therapy. The focus of this proposal is to identify mechanistic pathways to guide future therapeutic interventions for central sleep apnea based on the strong premise that multi-modality therapy will normalize respiration and hence mitigate adverse long-term consequences of CSA. The investigators' proposed studies will test combination therapies, including positive airway pressure (PAP) plus a pharmacological agent who have heart failure or are using opioid analgesics. The investigators anticipate that findings will inform future clinical trials to improve care and quality of life among Veterans suffering from central sleep apnea, which remains difficult to treat using existing approaches.

DETAILED DESCRIPTION:
All research activites are on hold due to COVID-19. We updated enrollment start date and we will update primary completion date and study completion date later.

This project is focused on identifying mechanistic pathways to guide future therapeutic interventions for central sleep apnea (CSA) based on the strong premise that multi-modality therapy - aiming to normalize respiration- is the requisite path to mitigating the long-term adverse consequences of CSA. The central hypothesis is that CSA reflects a combination of physiologic perturbations and may require combined modality therapy targeting different parts of the ventilatory feedback loop. The proposed studies will test combination therapies, including PAP plus a pharmacological agent. This will also increase the clinical relevance of the proposed studies since PAP therapy is typically prescribed as the initial treatment of CSA. To achieve the objectives of this proposal, the investigators will test the following three specific aims. Specific Aim (1) is to determine the effect of combination therapy aiming to dampen chemoreceptor sensitivity AND decreasing plant gain. The investigators hypothesize that combined therapy with PAP, acetazolamide and oxygen will be superior to each intervention alone in reducing central apnea-hypopnea index (CAHI) and the CO2 reserve during sleep in patients with central sleep apnea. Specific Aim (2) is to determine the effect of decreasing respiratory-related arousals on the propensity to develop central apnea. The investigators hypothesize that administration of PAP and zolpidem, will decrease respiratory-related arousals, CAHI and the CO2 reserve during sleep in patients with CSA compared to placebo. Specific Aim (3) is to determine the effect of augmenting serotonin A1 receptor activity on breathing during sleep. The investigators hypothesize that administration of PAP and buspirone, a serotonin A1 receptor agonist; will reduce the propensity to central apnea during sleep in Veterans with central sleep apnea. This Novel project seeks to identify physiologic pathways that can, in combination with PAP therapy, improve the effectiveness of treatment for patients with CSA. The proposed studies are innovative, feasible and will provide a much-needed roadmap for future clinical trials that are likely to transform the care of central apnea in Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Men and women Veterans with central sleep apnea, defined as Apnea Hypopnea Index (AHI)>15/hour with CAHI>5/hour, will be included in the experiments

Exclusion Criteria:

* less than 18 years old
* pregnant or breastfeeding female
* have severe respiratory disease that require to be on oxygen
* recent health event that may affect the ability to participate in the study,
* Body Mass Index (BMI) is >40 kg/m2
* significant insomnia
* mental instability
* recent health event that may affect sleep
* if at any time the principal investigator (PI) identifies that a certain drug is not suitable, or are unable to use the device that is used to treat sleep apnea, will be not be allowed to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CO2 reserve | 120 days
  CO2 reserve is the requisite change to induce central apnea is referred to as the CO2 reserve, which can be positive or negative.
Central apnea indices | 120 days
  Central apnea indices is used to indicate the severity of central sleep apnea

SECONDARY OUTCOMES:
Controller gain | 120 days
  Controller gain is a ventilatory response to changes in end-tidal PCO2
Plant gain | 120 days
  Plant gain is blood gas response to a change in ventilation. This measure represents the effectiveness of the "plant" in eliminating CO2.
Carotid body function | 120 days
  This measure represents the activity of the carotid bodies. It is measured by the decrease in ventilation in response to a single breath of 100% oxygen.
Peripheral chemoreflex sensitivity | 120 days
  Peripheral chemoreflex sensitivity is measured either via brief hypoxia or a single breath of CO2.
Respiratory arousal threshold | 120 days
  The nadir pressure in the upper airway (supra-glottic pressure) prior to the occurrence of an arousal.
% stable breathing | 120 days
  To assess breathing stability, the investigators will measure % stable breathing using minute ventilation (VE) and tidal volume (VT) coefficient of variation as indices of breathing instability.

CONTACTS AND LOCATIONS:
Overall Officials: M Safwan Badr, MD, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No